CLINICAL TRIAL: NCT01589042
Title: Chocolate Balloon Angioplasty Registry
Acronym: Chocolate BAR
Status: Completed | Type: Observational
Sponsor: TriReme Medical, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CLP782
Record Dates: First submitted 2012-04-27; First posted 2012-05-01 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Above the Knee: Patients treated with the Chocolate balloon for a lesion located above the knee
- Below the Knee: Patients treated with the Chocolate balloon for a lesion located below the knee

SUMMARY:
To collect data from real-world use with the Chocolate PTA Balloon Catheter to support the effectiveness of the device for use during percutaneous transluminal angioplasty (PTA) procedures.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years of age
2. Lesion successfully crossed with a guide-wire
3. Reference Vessel Diameter (RVD) within the treatment range of the Chocolate PTA Catheter used at the target lesion appropriate for 1:1 dilatation
4. Patient has given consent for their information to be submitted to this registry

Exclusion Criteria:

1. Lesion required stenting as the primary treatment approach
2. Life expectancy <12 months
3. Patient is enrolled in another clinical study that may impact the results of this registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Peripheral Arterial Disease appropriate for treatment with balloon angioplasty
Sampling Method: Non-Probability Sample
Enrollment: 490 (Actual)
Dates: Start 2012-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Achievement of Optimal PTA | average of 2 hours
  Percentage of PTA cases in which <30% diameter stenosis without a flow limiting dissection is achieved without the need for bail-out stenting

CONTACTS AND LOCATIONS:
Overall Officials: Jihad Mustapha, MD, Principal Investigator — Metro Health Hospital; Lawrence Garcia, MD, Principal Investigator — St Elizabeth's Med Center / Tufts Univ School of Medicine
Locations (13):
- United States (13):
  - Arizona Heart Institute, Phoenix, Arizona
  - Desert Cardiology, Rancho Mirage, California
  - Cardiovascular Research of North Florida, Gainesville, Florida
  - Mount Sinai Medical Center, Miami, Florida
  - Alexian Brothers Heart and Vascular, Elk Grove Village, Illinois
  - St. Elizabeth's Medical Center, Boston, Massachusetts
  - St. John's Hospital, Detroit, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Jackson Heart Clinic, Jackson, Mississippi
  - Rex Health, Raleigh, North Carolina
  - Cardiovascular Research of Dallas, Dallas, Texas
  - VA North Texas, Dallas, Texas
  - Wheaton Franciscan Healthcare, Racine, Wisconsin